CLINICAL TRIAL: NCT02677545
Title: Prevention of Cerebral Ischaemia in Stent Treatment for Carotid Artery Stenosis - A Randomised Multi-centre Phase II Trial Comparing Ticagrelor Versus Clopidogrel With Outcome Assessment on MRI (PRECISE-MRI)
Brief Title: Ticagrelor Versus Clopidogrel in Carotid Artery Stenting
Acronym: PRECISE-MRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5130C00171; me10Bonati
Record Dates: First submitted 2016-01-25; First posted 2016-02-09 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Ticagrelor; Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor & Aspirin (Experimental): Participants will receive a loading dose of 180 mg ticagrelor 1-3 days before stenting followed by a maintenance dose of 90 mg twice daily until 28-32 days after stenting. All participants will receive 75-100 mg aspirin per day throughout the study period.
  Interventions: Drug: Ticagrelor; Drug: Aspirin
- Clopidogrel & Aspirin (Active Comparator): Participants will receive a loading dose of 300 mg clopidogrel 1-3 days before stenting followed by a maintenance dose of 75 mg once daily until 28-32 days after stenting. All participants will receive 75-100 mg aspirin per day throughout the study period.
  Interventions: Drug: Clopidogrel; Drug: Aspirin

INTERVENTIONS:
Drug: Ticagrelor
  Other Names: Brilique
  Arms: Ticagrelor & Aspirin
Drug: Clopidogrel
  Other Names: Plavix
  Arms: Clopidogrel & Aspirin
Drug: Aspirin

SUMMARY:
Patients with symptomatic or asymptomatic carotid stenosis in whom carotid artery stenting is planned are randomised between antiplatelet therapy with ticagrelor plus aspirin or clopidogrel plus aspirin and examined with brain MRI before and after stent treatment. The proportion of patients with new ischaemic lesions on MRI after treatment is compared between the two groups.

DETAILED DESCRIPTION:
Carotid artery stenting (CAS) is an emerging treatment for atherosclerotic carotid stenosis. The main adverse event is embolic stroke during the procedure. Current medical management to prevent peri-procedural embolisation consists of dual antiplatelet therapy with clopidogrel and aspirin. Ticagrelor, a novel reversible inhibitor of the platelet adenosine diphosphate receptor P2Y12, was superior to clopidogrel, as add-on therapy to aspirin, in preventing stent thrombosis, cardiovascular outcome events, and death in patients undergoing coronary artery stenting, without causing an increase in major bleeding events. This study aims to test the hypothesis that ticagrelor is superior to clopidogrel as add-on to aspirin in preventing cerebral embolism during the CAS procedure.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent as documented by signature from the patient;
* Men or women ≥40 years of age;
* Moderate (50-69% narrowing of the artery according to the measuring method used in the NASCET trial64) or severe (70-99%) stenosis of the extracranial internal carotid artery caused by atherosclerosis;
* Symptomatic carotid stenosis (any transient or permanent symptoms caused by focal ischaemia in the vascular territory supplied by the carotid artery in the past 180 days, including ischaemic stroke, transient ischemic attack (TIA), amaurosis fugax or ischaemic retinal infarct), as long as the patient is clinically stable and able to walk unassisted (mRS ≤3) at the time of randomisation; or asymptomatic carotid stenosis (no ischaemic symptoms in the past 180 days);
* Stenosis amenable for treatment by CAS according to routine clinical work-up (degree of stenosis and suitability of vascular anatomy for CAS must be documented on vascular imaging within 90 days before the screening visit);
* CAS scheduled to take place within 1-3 days of randomisation.

Exclusion Criteria:

* Inability or unwillingness of the patient to understand and/or comply with study procedures and/or follow-up, e.g. due to language problems, psychological disorders, dementia, etc.;
* Women who are pregnant or breast feeding, or who intend to become pregnant during the course of the study. Women of childbearing age must take a blood pregnancy test to be eligible for the study within 14 days before randomisation;
* Lack of safe contraception, defined as: Female Participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the Investigator in individual cases. Female Participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential;
* Acute ischaemic stroke with symptom onset in the previous 24 hours before randomisation;
* atrial fibrillation;
* Fresh thrombus in the relevant carotid artery;
* Patient clinically unstable at the time of randomisation (includes worsening in NIH Stroke Scale of >2 points over the previous 24 hours);
* Patient unable to walk unassisted at the time of randomisation (mRS >3);
* Patients with known bleeding diathesis or coagulation disorder (e.g., thrombotic-thrombocytopenic purpura);
* Any active pathological bleed;
* Severe thrombocytopenia (platelet count <50'000/uL); platelet count must be documented within 30 days before randomisation
* History of previous symptomatic intracranial haemorrhage at any time (asymptomatic microbleeds do not qualify)
* History of gastrointestinal bleed within the past 6 months;
* Any contraindication to non-contrast MRI, including but not limited to: cardiac pacemaker incompatible with MRI; metal implants incompatible with MRI; claustrophobia);
* Contraindications to ticagrelor, clopidogrel, or acetylsalicylic acid (ASA), or to any of their excipients, including known hypersensitivity or allergy;
* Increased risk of bradycardic events (e.g., patients without a pacemaker who have sick sinus syndrome, 2nd or 3rd degree atrioventricular (AV) block, or history of bradycardia-related syncope; ECG must be obtained within 30 days before randomisation
* Need for medication not permitted during treatment period: Antithrombotic therapy other than Study Medication or permitted concomitant medication (see section 8.7) including: Antiplatelet therapy (other than ASA 100 mg daily), e.g.: open-label clopidogrel or ticagrelor; GPIIb/GPIIIa inhibitors, ticlopidine, prasugrel, dipyridamole, ozagrel, cilostazol; Therapeutic-dose anticoagulation (other than unfractioned heparin at the start of the CAS procedure), e.g.: phenprocoumon, warfarin, oral thrombin and factor Xa inhibitors, bivalirudin, hirudin, argatroban, unfractionated and low molecular weight heparins; Receipt of any intravenous or intra-arterial thrombolysis or mechanical thrombectomy within 24 hours prior to randomisation. If a patient requires intravenous or intra-arterial thrombolytic therapy during the treatment period, the Study Medication must be discontinued for at least 24 hours; Strong cytochrome P450 3A (CYP3A) inhibitors leading to substantial increases in ticagrelor plasma levels: ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin (but not erythromycin or azithromycin), nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir; or consumption of more than 1 litre of grapefruit juice daily; Strong CYP3A inducers leading to substantial decreases in ticagrelor plasma levels: rifampicin, rifabutin, phenytoin, carbamazepine, and phenobarbital; CYP3A substrates with narrow therapeutic indices which may be substantially increased by co-administration of ticagrelor: cyclosporine, quinidine, simvastatin at doses >40 mg daily or lovastatin at doses >40 mg daily. (Co-administration of ticagrelor with simvastatin increases simvastatin Cmax by 81% and area under curve (AUC) by 56% and increases simvastatin acid Cmax by 64% and AUC by 52% with some individual increases equal to 2- to 3-fold. Ticagrelor may have similar effect on lovastatin, but is not expected to have a clinically meaningful effect on other statins including atorvastatin and rosuvastatin); Anticipated requirement for long-term (>7 days) non-steroidal anti-inflammatory drugs (NSAIDs; short-term treatment with NSAIDs up to 7 days is allowed during the treatment period at the investigator's discretion);
* Need for any cardio-vascular surgery or cardio-vascular intervention other than the index CAS procedure for which the patient was randomised within the next 30 days after randomisation.
* Need for any other invasive procedure (surgery or intervention) other than the index CAS procedure for which the patient was randomised, which requires halting of Study Medication within the next 30 days after randomisation;
* History of major surgery within the past 30 days;
* Moderate or severe hepatic impairment;
* Renal impairment requiring dialysis;
* Known or suspected non-compliance, drug or alcohol abuse;
* Previous enrolment into the present study;
* Participation in another study with investigational drug within the 30 days preceding and during the present study;
* Patients incapable of judgment or patients under tutelage;
* Enrolment of the Investigator, his/her family members, employees and other dependent persons;

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
At least one new ischaemic brain lesion after CAS | Up to 32 days after CAS
  The primary efficacy outcome is the presence of at least one new ischaemic brain lesion on the second MRI scan done 1-3 days after CAS or on the third MRI scan done 28-32 days after CAS, which had not been present on the first MRI scan done 1-3 days before CAS.

SECONDARY OUTCOMES:
Composite of any stroke, myocardial infarction, major bleeding, or cardiovascular death | Through study completion, an average of 1 month after randomisation
  The clinical safety outcome is the composite of any stroke, myocardial infarction, major bleeding (including fatal, life-threatening or other major bleeding) or cardiovascular death occurring between randomisation and study completion.
Number of new ischaemic brain lesions after CAS | Up to 32 days after CAS
  A secondary efficacy outcome is the number of new ischaemic brain lesions on the second MRI scan done 1-3 days after CAS or on the third MRI scan done 28-32 days after CAS, which had not been present on the first MRI scan done 1-3 days before CAS.
Volume of new ischaemic brain lesions after CAS | Up to 32 days after CAS
  A secondary efficacy outcome is the total volume of new ischaemic brain lesions on the second MRI scan done 1-3 days after CAS or on the third MRI scan done 28-32 days after CAS, which had not been present on the first MRI scan done 1-3 days before CAS.
At least one new haemorrhagic brain lesion after CAS | Up to 32 days after CAS
  A secondary safety outcome is the presence of at least one new haemorrhagic brain lesion on the second MRI scan done 1-3 days after CAS or on the third MRI scan done 28-32 days after CAS, which had not been present on the first MRI scan done 1-3 days before CAS.

CONTACTS AND LOCATIONS:
Overall Officials: Leo H Bonati, MD, Principal Investigator — Department of Neurology and Stroke Center, University Hospital Basel
Locations (15):
- Belgium (2):
  - Ghent University Hospital - Dept thoracic and vascular surgery, Ghent
  - AZ Groeninge VZW, Kortrijk
- Germany (4):
  - University Hospital Aachen, Klinik für Diagnostische und Interventionelle Neuroradiologie, Aachen
  - Asklepios Kliniken Hamburg GmbH, Hamburg
  - Universitätsklinikum Heidelberg, Neurologische Klinik, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Kiel
- Italy (2):
  - Ospedale Civile di Mirano, Department of Cardiology, Mirano
  - UOC Neuroradiologia, Ospedale dell'Angelo, Venezia
- Netherlands (2):
  - AMC Medical Research BV on behalf of Academisch Medisch Centrum, Amsterdam
  - University Medical Center Utrecht, Utrecht
- Switzerland (4):
  - Kantonsspital Aarau Klinik für Neurologie, Aarau
  - University Hospital Basel, Basel
  - Insel Gruppe AG, Department of Neurology, Bern
  - Stadtspital Triemli Zürich/Department of Cardiology, Zurich
- Sheffield Clinical Research Facility, Northern General Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available for further analyses. Specific requests will be considered by the Trial Steering Committee.